CLINICAL TRIAL: NCT03818672
Title: Open Label Study to Evaluate the Steady-State Pharmacokinetics of Rifaximin 550 mg Tablets in Healthy Subjects and Subjects With Severe Hepatic Impairment
Brief Title: Steady-State Pharmacokinetics of Rifaximin 550 mg Tablets in Healthy and Hepatically Impaired Subjects
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study determined to be infeasible.
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RFPK4045
Record Dates: First submitted 2019-01-22; First posted 2019-01-28 (Actual); Results first posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Severe Hepatic Impairment
MeSH Terms: interventions — Rifaximin

STUDY DESIGN:
Intervention Model Description: open-label, repeat-dose, parallel-design study in 12 subjects with severe hepatic impairment and 6 healthy subjects with normal hepatic function.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rifaximin (Experimental): Rifaximin 550 mg BID
  Interventions: Drug: Rifaximin

INTERVENTIONS:
Drug: Rifaximin — Rifaximin 550 MG BID

SUMMARY:
The primary objective of this study is to characterize the steady state plasma

DETAILED DESCRIPTION:
The primary objective of this study is to characterize the steady state plasma PK of rifaximin (550 mg BID) in subjects with severe hepatic impairment (MELD 19 to 25 and MELD >25), as well as healthy subjects with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

* Hepatically impaired subjects will be ≥18 years of age, have a diagnosis of liver cirrhosis and a MELD score of ≥19 at Screening. Note: At least 6 of the hepatically impaired subjects will have a MELD score of >25.

Exclusion Criteria:

* Subject has known allergy to rifaximin, rifampin, or other rifamycins, excipients and/or vehicles used in the formulation, or any other clinically significant allergies.
* Subject has participated in an investigational drug or device study within 30 days prior to Day 1 (Baseline).
* Subject has any concurrent illness (other than liver cirrhosis), disability or circumstance that may affect the interpretation of clinical data, could cause noncompliance with treatment or visits or otherwise contraindicates participation in this study in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2020-02-02 (Actual); Study Completion 2020-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Varsha Bhatt, Study Director — Bausch Health Companies
Locations (1):
- Valeant Site 01, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rifaximin
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Rifaximin
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (6.870)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Model for End Stage Liver Disease Score at baseline: Healthy [Count of Participants; unit: Participants] — MELD score was calculated based on laboratory results using the following formula:
  • (0.957 * ln(Serum Creatinine mg/dL) + 0.378 * ln(Serum Bilirubin mg/dL) + 1.120 * ln( international normalised ratio [INR] blood test ) + 0.643) * 10.
  Participants | 1
Model for End Stage Liver Disease Score at baseline: 19 to 25 [Count of Participants; unit: Participants] — MELD score was calculated based on laboratory results using the following formula:
  • (0.957 * ln(Serum Creatinine mg/dL) + 0.378 * ln(Serum Bilirubin mg/dL) + 1.120 * ln( international normalised ratio [INR] blood test ) + 0.643) * 10.
  Participants | 4

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: Maximum observed plasma concentration (Cmax) of rifaximin and 25-desacetyl rifaximin, if measurable
Time Frame: 7 days
Population: Participants with Model for End Stage Liver Disease (MELD) of 19 to 25 (N=4) were assessed for pharmacokinetic parameters. There were too few healthy participants (N=1) to assess.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Rifaximin
Number analyzed (Participants) | 4
ng/mL
  rifaximin | 13.4 (90.0)
  25-desacetyl rifaximin | 0.356 (87.5)

2. Primary Outcome: Time of the Maximum Concentration (Tmax)
Description: Time of the maximum concentration (Tmax) of rifaximin and 25-desacetyl rifaximin, if measurable
Time Frame: 7 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Rifaximin
Number analyzed (Participants) | 4
hours
  rifaximin | 0.688 (0.688)
  25-desacetyl rifaximin | 0.625 (0.750)

3. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) During the 12-hour Dose Interval
Description: Area under the plasma concentration versus time curve (AUC) during the 12-hour dose interval of rifaximin and 25-desacetyl rifaximin, if measurable
Time Frame: 7 days
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Rifaximin
Number analyzed (Participants) | 4
h*ng/mL
  rifaximin | 98.7 (107)
  25-desacetyl rifaximin | 3.04 (85.2)

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Rifaximin
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 2/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rifaximin (N=5)
Vomiting (Gastrointestinal disorders) | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor for details.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-08): https://cdn.clinicaltrials.gov/large-docs/72/NCT03818672/Prot_SAP_000.pdf